CLINICAL TRIAL: NCT00663026
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Safety, Tolerability, Reactogenicity, And Pharmacokinetic Study Of Bapineuzumab (AAB 001) Administered Subcutaneously In Subjects With Mild To Moderate AD
Brief Title: Study Evaluating Bapineuzumab In Alzheimer Disease Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3133L1-2203; B2521008
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-09

CONDITIONS: Alzheimer Disease
Keywords: antibody; immunotherapy
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): 5 mg/week
  Interventions: Drug: bapineuzumab
- B (Experimental): 10 mg/week
  Interventions: Drug: bapineuzumab
- C (Experimental): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bapineuzumab — 5 mg bapineuzumab subcutaneous injection once per week for 6 months
  Arms: A
Drug: bapineuzumab — 10 mg bapineuzumab subcutaneous injection once per week for 6 months
  Arms: B
Drug: placebo — Placebo subcutaneous injection once per week for 6 months
  Arms: C

SUMMARY:
The study will evaluate the safety and effectiveness of bapineuzumab for the treatment of mild to moderate Alzheimer disease. Subjects will be in the study for six months and will receive subcutaneous injections once per week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer Disease according to National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria
* Mini-Mental State Examination (MMSE) score 16-26

Exclusion Criteria:

* Magnetic Resonance Imaging (MRI) showing other brain abnormalities
* Other diagnosed neurological or psychiatric disorders

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (17):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Los Alamitos, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Delray Beach, Florida
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Lawrenceville, Georgia
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, East Providence, Rhode Island
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Bennington, Vermont
  - Pfizer Investigational Site, Madison, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3133L1-2203&StudyName=Study%20Evaluating%20Bapineuzumab%20In%20Alzheimer%20Disease%20Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo matched to bapineuzumab subcutaneous injection once weekly for 6 months.
- Bapineuzumab 5 mg: Bapineuzumab 5 milligram (mg) subcutaneous injection once weekly for 6 months.
- Bapineuzumab 10 mg: Bapineuzumab 10 mg subcutaneous injection once weekly for 6 months.
Period: Overall Study
Arm/Group | Placebo | Bapineuzumab 5 mg | Bapineuzumab 10 mg
Started | 19 | 29 | 31
Completed | 17 | 23 | 27
Not Completed | 2 | 6 | 4
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other | 1 | 2 | 0
Not completed — Adverse Event | 0 | 2 | 3
Not completed — Caregiver Request | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bapineuzumab 5 mg | Bapineuzumab 10 mg | Total
Number analyzed (Participants) | 19 | 29 | 31 | 79
Age Continuous [Mean (Standard Deviation); unit: years] | 76.16 (8.63) | 71.28 (8.73) | 72.42 (8.83) | 72.90 (8.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 18 | 12 | 38
  Male | 11 | 11 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 30 days after Week 25 dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline up to 30 days after Week 25 dose
Population: Safety population included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Bapineuzumab 5 mg | Bapineuzumab 10 mg
Number analyzed (Participants) | 19 | 29 | 31
participants
  AEs | 16 | 22 | 28
  SAEs | 1 | 2 | 3

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Time Frame: Predose, 4 hours [hrs] postdose, 72 hrs postdose on Day 3 of Week 0 and 25; Predose on Day 7 (Week 1), Week 10, 14, 16, 18, 22, 26, 30; Predose and 4 hrs postdose on Week 12
Population: Pharmacokinetic (PK) analysis set included all participants who provided data for the estimation of at least 1 of the relevant PK parameters (Cmax, time to maximum concentration [tmax], area under the curve [AUC], terminal elimination half-life [t1/2], apparent systemic clearance [CL/F], and apparent volume of distribution [Vz/F]).
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Bapineuzumab 5 mg | Bapineuzumab 10 mg
Number analyzed (Participants) | 29 | 31
nanogram per milliliter (ng/mL) | 4219.97 (945.23) | 8012.88 (2793.53)

3. Secondary Outcome: Average Serum Concentration at Steady State (Cavg,ss)
Description: Average plasma concentration at steady state (Cavg,ss) = AUCtau divided by dosing interval (1 week). AUCtau is the area under the plasma concentration time curve (AUC) at steady state from time zero (pre-dose) to end of dosing interval (tau), here dosing interval is 1 week.
Time Frame: Predose, 4 hrs postdose, 72 hrs postdose on Day 3 of Week 0 and 25; Predose on Day 7 (Week 1), Week 10, 14, 16, 18, 22, 26, 30; Predose and 4 hrs postdose on Week 12
Population: PK analysis set included all participants who provided data for the estimation of at least 1 of the relevant PK parameters (Cmax, tmax, AUC, t1/2, CL/F and Vz/F). Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bapineuzumab 5 mg | Bapineuzumab 10 mg
Number analyzed (Participants) | 25 | 29
ng/mL | 3123.071 (1074.116) | 6912.301 (2149.143)

4. Secondary Outcome: Serum Decay Half-Life (t1/2)
Description: Serum decay half-life is the time measured for the serum concentration to decrease by one half.
Time Frame: as for outcome 3
Population: t1/2 not calculated due to inadequate characterization of the terminal elimination phase.
Arm/Group | Bapineuzumab 5 mg | Bapineuzumab 10 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax)
Time Frame: as for outcome 3
Population: PK analysis set included all participants who provided data for the estimation of at least 1 of the relevant PK parameters (Cmax, tmax, AUC, t1/2, CL/F and Vz/F).
Measure: Median (Full Range); unit: hours
Arm/Group | Bapineuzumab 5 mg | Bapineuzumab 10 mg
Number analyzed (Participants) | 29 | 31
hours | 3696.00 [1680.00 to 4368.00] | 4200.00 [72.00 to 4368.00]

6. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau)
Description: AUCtau is the area under the serum concentration time curve (AUC) at steady state from time zero (pre-dose) to end of dosing interval (tau), here dosing interval is 1 week.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Bapineuzumab 5 mg | Bapineuzumab 10 mg
Number analyzed (Participants) | 25 | 31
ng*hr/mL | 524675.88 (180451.56) | 1161266.63 (361056.04)

7. Secondary Outcome: Apparent Systemic Clearance (CL/F)
Description: Clearance (CL) of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after subcutaneous dose (apparent systemic clearance) is influenced by the fraction (F) of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Steady-state apparent systemic clearance (CL/F) was calculated as dose/AUC tau.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milliliter/hour/kilogram (mL/hr/kg)
Arm/Group | Bapineuzumab 5 mg | Bapineuzumab 10 mg
Number analyzed (Participants) | 25 | 29
milliliter/hour/kilogram (mL/hr/kg) | 0.16 (0.05) | 0.132 (0.069)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Bapineuzumab 5 mg | Bapineuzumab 10 mg
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/29 | 3/31
Other Adverse Events (participants affected / at risk) | 15/19 | 22/29 | 27/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Bapineuzumab 5 mg (N=29) | Bapineuzumab 10 mg (N=31)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Serum sickness (Immune system disorders) | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0
Subdural hemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | Bapineuzumab 5 mg (N=29) | Bapineuzumab 10 mg (N=31)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Fatigue (General disorders) | 2 | 2 | 0
Injection site erythema (General disorders) | 1 | 2 | 1
Injection site haemorrhage (General disorders) | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 6
Urinary tract infection (Infections and infestations) | 2 | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Atypical fibroxanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 2 | 2
Headache (Nervous system disorders) | 2 | 2 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 2 | 6
Agitation (Psychiatric disorders) | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Designation of outcomes as primary, secondary was based on study team's input as study did not specify them as primary or secondary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.